CLINICAL TRIAL: NCT07205146
Title: Evolution of Symptoms After Treatment With System CavatermTM for Idiopathic Functional Menometrorraghia Contraceptive Implants
Brief Title: CavatermTM for Idiopathic Functional Menometrorraghia
Acronym: CAVATERM
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 25-5206
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Cavaterm™ System
Keywords: Cavaterm™ system; idiopathic functional menometrorrhagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cavaterm: patients who received treatment with the Cavaterm™ system for idiopathic functional menometrorrhagia
  Interventions: Other: menometrorrhagia

INTERVENTIONS:
Other: menometrorrhagia — rate of menometrorrhagia at 2 months after treatment

SUMMARY:
The prevalence of menometrorrhagia is estimated at 11% to 13% in the general population and increases with age to reach 24% in 36-40 year olds. It is the leading cause of gynecological consultations. Considered benign, menometrorrhagia is responsible for anemia and impaired quality of life. It is the most common cause of iron deficiency anemia in premenopausal women.

The etiology of menometrorrhagia is varied. The main causes of menometrorrhagia are organic causes, iatrogenic causes, coagulopathies, hypothyroidism, and endometrial atrophy. In the majority of cases, no underlying pathology is found; they are then called functional idiopathic. This is a diagnosis of exclusion.

In idiopathic functional menometrorrhagia, the first-line treatment is medical. In the event of failure of medical treatment (in 50% of cases), in women who do not wish to maintain their reproductive possibilities, surgical treatment may be considered.

The Cavaterm™ system is a balloon-assisted endometrial ablation device. Treatment with Cavaterm™ involves removing the endometrium using a minimally invasive technique. The procedure is short-term and outpatient.

In this study, we aim to evaluate the Cavaterm™ system for the treatment of idiopathic functional menometrorrhagia.

ELIGIBILITY:
* Inclusion Criteria * :

  * women over 18
  * patient who benefited from treatment with the Cavaterm™ system for idiopathic functional menometrorrhagia
  * treatment between January 2024 and December 2024
  * person having expressed his non-opposition
* Exclusion Criteria * :

  * inability to understand the information given
  * person deprived of liberty
  * person under guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This study includes all patients who received treatment with the Cavaterm™ system for idiopathic functional menometrorrhagia between January 2024 and December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
menometrorrhagia | at 2 months after treatment
  rate of menometrorrhagia at 2 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mère Enfant, Lyon, France